CLINICAL TRIAL: NCT02187692
Title: The Effectiveness of The Meta-cognitive Training Among Chronic Schizophrenia Patients Treated Within Community Support Groups in Poland.
Brief Title: The Effectiveness of the Meta-cognitive Training Among Patients With Chronic Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Gawęda, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCTPOLAND
Record Dates: First submitted 2013-10-14; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia;; meta-cognition;; general functioning;; positive symptoms;; insight;
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU (No Intervention): Treatment as Usual (TAU) vs meta-cogntive training (MCT) condition will be contrasted. In the TAU patients attend regular day programm that includes psychoeducation, social training, vocational rehabilitation, psychotherapy. The MCT condition is an active condition that includes structuralized therapy modules twice a week for four weeks (eight modules in total). There will be no additional differences in the interventions between two groups. Participants will be randomized from patients from the same population into two conditions.
- MCT (Experimental): Treatment as Usual (TAU) vs meta-cogntive training (MCT) condition will be contrasted. In the TAU patients attend regular day programm that includes psychoeducation, social training, vocational rehabilitation, psychotherapy. The MCT condition is an active condition that includes structuralized therapy modules twice a week for four weeks (eight modules in total). There will be no additional differences in the interventions between two groups. Participants will be randomized from patients from the same population into two conditions.
  Interventions: Behavioral: MCT

INTERVENTIONS:
Behavioral: MCT — The meta-cognitive training (the MCT) consists of eight structurized psychological therapy modules that provides basic knowledge about cognitive biases that are associated with schizophrenia and it provides the sklills how to overcome negative consequences of the biases. The MCT includes: Module 1 manages self-serving bias (i.e. external-personal attribution for failure, internal attribution for positive events); Module 2 and 7 target the jumping to conclusion; Module 3 and 7 concern beliefs flexibility and bias against disconfirmatory evidence; Module 4 and 6 target deficits in theory of mind; Module 5 is devote to ameliorate the cognitive over-confidence in false memories; Module 8 deals with depressive thinking style.
  Arms: MCT

SUMMARY:
The aim of the study is to compare the effectiveness of the meta-cognitive training (MCT) for schizophrenia against treatment as usual (TAU) among patients who attends community support groups. 4 weeks of MCT will be administered for patients two times per week. MCT consists of well structured cognitive behavioral therapy interventions. MCT will be administered according authors recommendations. All participants will be assessed at baseline (T0) and up to one week after the MCT intervention (T1, 4-5 week of the study).

DETAILED DESCRIPTION:
50 patients with established schizophrenia diagnosis will be included and randomized into two conditions: MCT (n= 25) and TAU (n=25). Exclusion criteria are: neurological diseases, substance dependence (alcohol and drugs).

A broad outcome measures will be provided including symptoms severity, cognitive biases, neurocognition, insight and social functioning. Changes in variable after the intervention will be compared between two condition.

Only patients with established schizophrenia with no neurological diseases will be included.

All patients will be assessed at two time points: T0 - at baseline, up to one week before the intervention starts and T1 up to one week after the intervention is finished. T1 assessment will be at 4-5 weeks after the study begun.

Measures

1. General functioning General Assessment of Functioning was used as a measure of the severity of patients' functional disabilities.
2. Insigh A questionnaire of insight into schizophrenia consists of six items targeting insight. The scale has a good reliability with Cronbach's alpha 0.8.
3. The subjective sense of influence on the course of schizophrenia The Brief Measure to Assess Perception of the Self-influence on the Disease Course - Version for Schizophrenia consists of five items targeting different aspects of subjective sense of influence on the course of schizophrenia. The scale has satisfactory psychometric properties (Cronbach's alpha= 0.78).

4, Psychotic symptoms The severity of delusions and hallucinations were assessed at the baseline and after the intervention with the semi-structured Psychotic Symptom Rating Scale (The PSYRATS). The PSYRATS comprises hallucination and delusions subscale, each design to assess psychological aspects of the symptoms on a five point scale from 0 to 4. The items for the hallucination scale are: frequency (PH1); duration (PH2); location (PH3); loudness (PH4); beliefs regarding the origin of voices (PH5); amount of negative content of voices (PH6); degree of negative content (PH7); amount of distress (PH8); intensity of distress (PH9); disruption to life caused by voices (PH10); controlability of voices (PH11). The delusion subscale consists of six items: amount of preoccupation with delusions (PD1); duration of preoccupation with delusions (PD2); conviction (PD3); amount of distress (PD4); intensity of distress (PD5); disruption to life caused by beliefs (PD6). The PSYRATS has good psychometric properties and have been reported being sensitive to symptoms change over time. In addition the Paranoia Checklist which comprises 18 items, each rated on 5 point scale for frequency, distress and degree of conviction, was used in order to assess delusional ideations. The participants were asked to state if they experience different delusional ideation during the last week before filling out the questionnaire.

5. Cognitive Biases. Cognitive Biases Questionnaire for Psychosis consists of 30 vignettes of everyday life scenarios. Participants are asked to imagine themselves as being in the situation and then choose one out of four cognitive responses indicating specific cognitive biases. CBQp comprises of seven subscales: anomalous perceptions (AP); threatening events (TE); intentionalising (I); catastrophising (C); dichotomous thinking (DT); jumping to conclusion (JTC); emotion based reasoning (ER).

In addition two behavioral tasks were used in order to assess the most prominent cognitive biases in schizophrenia, that is to say jumping to conclusion and theory of mind deficits. In the Fish Task the participants are presented with two lakes with different proportion of grey and orange fishes. In the first lake (lake A) there is 80% grey and 20% of orange fishes. The proportion of fishes in the lake B is reversed. Participants are presented with the fisherman who stands between lakes to catch fishes, but he is allowed to do that only from one lake during the entire experiment. Participants on the computer screen were presented with fishes. Two responses were gathered: 1) the participant should make the confidence judgment by indicating from 0-100% how confident they are regarding the fish is from lake A or lake B; 2) whether the participant has enough evidences for the final decision on the fish is from lake A or B. Two alternative versions of the Fish Task were used for pre- and post-test. We analyzed a number of fishes that were considered by participants for the final decision. The less fishes were considered the more the participant has jumping to conclusions tendencies.

Reading the Mind from Eyes Test (RMET,) was used in order to assess the deficits in the theory of mind. The test consists of 36 different faces pictures restricted to eyes area only. Based on the face expression participant is asked to infer the emotional state of the person presented on the picture. We split the original 36 pictures test into two separate tests for the pre- and post-test. In addition to original test we included the conviction question in which participants responded how confident they are in their decisions (100% sure). The RMET test has good psychometric properties and has been used often in schizophrenia.

6. Global neurocognitive functioning Trial making test (TMT) A and B was used to assess global cognitive flexibility. TMT A test is design to test psychomotor speed and attention. TMT B test targets the data on the cognitive flexibility.

All tests will be administered at T0 (baseline assessment up to one week before intervention) and T1 (up to one week after the intervention ).

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia diagnosis accotding to the ICD-10 criteria
* attending local community support groups for psychitatric patients

Exclusion Criteria:

* neurological diseases
* substance abuse
* severe psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptom Rating Scale (The PSYRATS) | week 0
  The severity of delusions and hallucinations were assessed at the baseline and after the intervention with the semi-structured Psychotic Symptom Rating Scale. The PSYRATS comprises hallucination and delusions subscale, each design to assess psychological aspects of the symptoms on a five point scale from 0 to 4.
[change] Psychotic Symptom Rating Scale (The PSYRATS) | week 4-5
  The severity of delusions and hallucinations were assessed at the baseline and after the intervention with the semi-structured Psychotic Symptom Rating Scale. The PSYRATS comprises hallucination and delusions subscale, each design to assess psychological aspects of the symptoms on a five point scale from 0 to 4.

SECONDARY OUTCOMES:
Cognitive Biases Questionnairre for Psychosis (CBQp) | week 0
  Cognitive Biases Questionnaire for Psychosis (CBQp) consists of 30 vignettes of everyday life scenarios. Participants are asked to imagine themselves as being in the situation and then choose one out of four cognitive responses indicating specific cognitive biases. CBQp comprises of seven subscales: anomalous perceptions (AP); threatening events (TE); intentionalising (I); catastrophising (C); dichotomous thinking (DT); jumping to conclusion (JTC); emotion based reasoning (ER).
[Change] Cognitive Biases Questionnairre for Psychosis (CBQp) | week 4-5
  Cognitive Biases Questionnaire for Psychosis (CBQp) consists of 30 vignettes of everyday life scenarios. Participants are asked to imagine themselves as being in the situation and then choose one out of four cognitive responses indicating specific cognitive biases. CBQp comprises of seven subscales: anomalous perceptions (AP); threatening events (TE); intentionalising (I); catastrophising (C); dichotomous thinking (DT); jumping to conclusion (JTC); emotion based reasoning (ER).

OTHER OUTCOMES:
Neurocognition | week 0
  Trial making test (TMT) A and B was used to assess global cognitive flexibility. TMT A test is design to test psychomotor speed and attention. TMT B test targets the data on the cognitive flexibility.
[Change] Neurocognition | week 4-5
  Trial making test (TMT) A and B was used to assess global cognitive flexibility. TMT A test is design to test psychomotor speed and attention. TMT B test targets the data on the cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Gawęda, PhD, Principal Investigator — II Department of Psychiatry, Medical University of Warsaw
Locations (1):
- II Department of Psychiatry, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Gaweda L, Krezolek M, Olbrys J, Turska A, Kokoszka A. Decreasing self-reported cognitive biases and increasing clinical insight through meta-cognitive training in patients with chronic schizophrenia. J Behav Ther Exp Psychiatry. 2015 Sep;48:98-104. doi: 10.1016/j.jbtep.2015.02.002. Epub 2015 Mar 5. PMID 25775947